CLINICAL TRIAL: NCT03491046
Title: Molecular Imaging Assessment of ACL Viability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP0649/2013H0009
Record Dates: First submitted 2018-03-30; First posted 2018-04-09 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patient population with ACL injury or reconstruction (Experimental)
  Interventions: Device: PET scan; Device: MRI scan
- Patient population without ACL injury or reconstruction (Experimental)
  Interventions: Device: PET scan; Device: MRI scan

INTERVENTIONS:
Device: PET scan — low dose fluorodeoxyglucose (FDG) PET research scan with CEST sequence
Device: MRI scan — standard of care MRI

SUMMARY:
The objective of this study is to answer the following questions:

1. Does the appearance of the reconstructed anterior cruciate ligament (ACL) vary in appearance on PET/MRI depending on graft type and time after surgery?
2. What is the appearance of the native ACL on Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI)?

DETAILED DESCRIPTION:
This Phase I feasibility trial will evaluate knee injuries utilizing a standard of care non-contrast 3 Tesla (T) MRI. In addition, knee injuries will be assessed with a low dose (1/5 of the dose given for standard of care PET scans) fluorodeoxyglucose (FDG) PET research scan with CEST sequences. Patients enrolled in this study will include both those with and without a history of ACL repair; however, patients receiving the standard of care MRI will not be currently suspected of having an ACL injury based on physical examination and history.

Patients with and without a history of ACL reconstruction will undergo a low dose FDG PET scan in the same setting as their MRI. The PET examination will be performed such that the early phase of imaging is performed prior to the MRI and the delayed phase is completed immediately following the MRI. This dual-phase scanning will allow for both assessment of the vascularity of the graft as well as its metabolic activity.

Patients will be asked to provide study personnel with authorization to their medical records regarding the outcome of the knee graft. This authorization will be provided for 10 years from date of signed consent.

Comparisons of the finding in normal and reconstructed ligaments as well as between graft types based on time from reconstruction will demonstrate the feasibility of this imaging technique and allow for generation of an imaging based hypothesis that will provide metabolic activity of the graft in a post-operative knee.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 60 years of age.
* Patients scheduled for a standard of care MRI at OSU.

Exclusion Criteria:

* Patients with a suspected ACL injury.
* Patients who are pregnant or lactating.
* Patients who are prisoners.
* Patients who are unable to provide consent.
* Patient with significant renal insufficiency, i.e. an estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73m2.
* Patients who exhibit noticeable anxiety and/or claustrophobia or who exhibit sever vertigo when they are moved into the MR.
* Subjects with any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc.).
* Subjects with any type of ferromagnetic bioimplant that could potentially be displaced or damaged.
* Subjects that have vascular or aneurysm clips, or metallic staples from a surgical procedure.
* Subjects with permanent tattoo eye liner (may contain metallic coloring).
* Subjects that may have shrapnel imbedded in their bodies, such as from war wounds, metal workers and machinists (metallic fragments in or near eyes), severe auto accident victims.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
metabolic activity in the ACL graft | through study completion, an average of 2-5 years
  We will assess the metabolic activity in the ACL graft by measuring the maximum standard uptake value of the PET signal within the graft, bone tunnels, and surrounding healthy tissue.
feasibility of imaging | through study completion, an average of 2-5 years
  We will determine the feasibility of imaging ACL grafts using FDG PET/CT by performing imaging in a variety of patients, with different surgical techniques and times since surgery. Whether a sufficiently measurable signal is achieved will be evaluated alongside the signal in the healthy, control knee of each patient.
the ability of coregistration of PET and MR | through study completion, an average of 2-5 years
  We will evaluate the ability to coregister separately acquired PET and MR images by creating a foam mold of the MRI knee coil to be used as a positioning device during the separate PET/CT imaging. We will assess the impact of motion artifacts on both image data sets as well.
dynamic uptake rate of FDG in the ACL graft | through study completion, an average of 2-5 years
  The PET images will be acquired in a dynamic mode, meaning they can be reconstructed into frames of different durations over the total 75 minute scan time. We will assess the uptake at the end of the 75 minute imaging period, as well as the dynamic uptake rate of FDG in the ACL graft, to learn whether the rate of uptake can provide additional insight into the healing process.

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2013-03-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03491046/Prot_000.pdf